CLINICAL TRIAL: NCT04789499
Title: Smell in Covid-19 and Efficacy of Nasal Theophylline
Acronym: SCENT2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202101190
Record Dates: First submitted 2021-03-08; First posted 2021-03-09 (Actual); Results first posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-04

CONDITIONS: Covid19; Anosmia; Olfactory Disorder; Covid-19 Pandemic; SARS-CoV-2 Infection; Hyposmia; Ageusia; Hypogeusia
Keywords: Smell; Smell loss; smell dysfunction; olfactory dysfunction; COVID-19; anosmia; theophylline; nasal irrigation
MeSH Terms: conditions — COVID-19; Anosmia; Ageusia; Olfaction Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The pharmacy will maintain the blind until the completion of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Theophylline (Experimental): 400mg theophylline capsule diluted in 240 mL isotonic nasal saline lavage twice daily for six weeks.
  Interventions: Drug: Theophylline Powder
- Placebo (Placebo Comparator): 500mg lactose capsule diluted in 240 mL isotonic nasal saline lavage twice daily for six weeks.
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: Theophylline Powder — Twice daily nasal irrigation with 400 mg theophylline capsules and USP Grade Sodium Chloride & Sodium Bicarbonate Mixture (pH balanced, Isotonic & Preservative & Iodine Free) commercially prepared packets dissolved in 240 ml of distilled water.
  Other Names: Theophylline nasal irrigation
  Arms: Theophylline
Drug: Placebo Comparator — Twice daily nasal irrigation with 500 mg lactose powder capsules and USP Grade Sodium Chloride & Sodium Bicarbonate Mixture (pH balanced, Isotonic & Preservative & Iodine Free) commercially prepared packets dissolved in 240 ml of distilled water.
  Other Names: lactose powder
  Arms: Placebo

SUMMARY:
Evidence of COVID-19 related anosmia and dysgeusia continues to accumulate daily.

Currently, up to 80% of patients report subjective olfactory dysfunction (OD), and prevalence using objective olfactory testing could be even higher.

We propose a phase II single-site, double-blinded, placebo-controlled randomized clinical trial to determine the efficacy and safety of intranasal theophylline, a known phosphodiesterase inhibitor in the treatment of asthma, as a possible treatment for COVID-19 related OD. Theophylline has shown benefit in similar clinical trials for post-viral OD.

DETAILED DESCRIPTION:
Post-viral olfactory dysfunction has numerous known adverse effects such as loss of cortical gray matter and decrease in quality of life. COVID-19 related olfactory dysfunction has already been shown to be correlated with depression and decreased quality of life, so finding an effective treatment is imperative.

Intranasal and oral corticosteroids as well as olfactory training are currently used to treat post-viral OD; however they have demonstrated limited efficacy and there is no current gold standard of care. There is no current consensus on the pathogenesis of COVID-related anosmia; however evidence for post-viral olfactory dysfunction suggests sensory axonal regeneration and olfactory signaling may rely on elevated levels of secondary messengers cAMP and cGMP, a known effect of theophylline. In this phase II treatment trial, patients will be allocated 1:1 to receive either intranasal theophylline irrigation or placebo for six weeks. Various smell surveys and scratch-and-sniff tests will be utilized to capture changes in smell ability.

Due to COVID-19, this study will be conducted virtually, except for the first ten enrolled patients who will undergo one serum theophylline test. This study is limited to patients living in Missouri or Illinois.

ELIGIBILITY:
Inclusion Criteria:

* Olfactory dysfunction that has persisted for >3 months following suspected COVID-19 infection
* Residing within the states of Missouri or Illinois.
* Can read, write, and understand English.

Exclusion Criteria:

* History of olfactory dysfunction prior to COVID-19 infection
* Use of concomitant therapies specifically for the treatment of olfactory dysfunction
* History of olfactory dysfunction longer than 12 months
* Known existence of nasal polyps, prior sinonasal, or anterior skull-based surgery
* Dependence on theophylline for comorbid conditions such as asthma and COPD
* History of an allergic reaction to theophylline or other methylxanthines
* History of neurodegenerative disease (ie. Alzheimer's dementia, Parkinson's disease, Lewy body dementia, frontotemporal dementia)
* Pregnant or breastfeeding mothers
* Current use of medications with significant interactions with theophylline, which include cimetidine, ciprofloxacin, disulfiram, enoxacin, fluvoxamine, interferon-alpha, lithium, mexiletine, phenytoin, propafenone, propranolol, tacrine, thiabendazole, ticlopidine, and troleandomycin.
* Pre-existing arrhythmias or seizures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay F Piccirillo, M.D., FACS, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine in Saint Louis, St Louis, Missouri, United States

REFERENCES:
- [Background] Khan AM, Kallogjeri D, Piccirillo JF. Growing Public Health Concern of COVID-19 Chronic Olfactory Dysfunction. JAMA Otolaryngol Head Neck Surg. 2022 Jan 1;148(1):81-82. doi: 10.1001/jamaoto.2021.3379. PMID 34792577
- [Background] Hoffman HJ, Rawal S, Li CM, Duffy VB. New chemosensory component in the U.S. National Health and Nutrition Examination Survey (NHANES): first-year results for measured olfactory dysfunction. Rev Endocr Metab Disord. 2016 Jun;17(2):221-40. doi: 10.1007/s11154-016-9364-1. PMID 27287364
- [Background] Whitcroft KL, Hummel T. Olfactory Dysfunction in COVID-19: Diagnosis and Management. JAMA. 2020 Jun 23;323(24):2512-2514. doi: 10.1001/jama.2020.8391. No abstract available. PMID 32432682
- [Background] Speth MM, Singer-Cornelius T, Oberle M, Gengler I, Brockmeier SJ, Sedaghat AR. Mood, Anxiety and Olfactory Dysfunction in COVID-19: Evidence of Central Nervous System Involvement? Laryngoscope. 2020 Nov;130(11):2520-2525. doi: 10.1002/lary.28964. Epub 2020 Aug 12. PMID 32617983
- [Background] Burges Watson DL, Campbell M, Hopkins C, Smith B, Kelly C, Deary V. Altered smell and taste: Anosmia, parosmia and the impact of long Covid-19. PLoS One. 2021 Sep 24;16(9):e0256998. doi: 10.1371/journal.pone.0256998. eCollection 2021. PMID 34559820
- [Background] Schiffman SS, Warwick ZS. Flavor enhancement of foods for the elderly can reverse anorexia. Neurobiol Aging. 1988 Jan-Feb;9(1):24-6. doi: 10.1016/s0197-4580(88)80009-5. PMID 3164095
- [Background] Murphy C, Schubert CR, Cruickshanks KJ, Klein BE, Klein R, Nondahl DM. Prevalence of olfactory impairment in older adults. JAMA. 2002 Nov 13;288(18):2307-12. doi: 10.1001/jama.288.18.2307. PMID 12425708
- [Background] Bitter T, Gudziol H, Burmeister HP, Mentzel HJ, Guntinas-Lichius O, Gaser C. Anosmia leads to a loss of gray matter in cortical brain areas. Chem Senses. 2010 Jun;35(5):407-15. doi: 10.1093/chemse/bjq028. Epub 2010 Mar 15. PMID 20231262
- [Background] Pinto JM, Wroblewski KE, Kern DW, Schumm LP, McClintock MK. Olfactory dysfunction predicts 5-year mortality in older adults. PLoS One. 2014 Oct 1;9(10):e107541. doi: 10.1371/journal.pone.0107541. eCollection 2014. PMID 25271633
- [Background] Liu B, Luo Z, Pinto JM, Shiroma EJ, Tranah GJ, Wirdefeldt K, Fang F, Harris TB, Chen H. Relationship Between Poor Olfaction and Mortality Among Community-Dwelling Older Adults: A Cohort Study. Ann Intern Med. 2019 May 21;170(10):673-681. doi: 10.7326/M18-0775. Epub 2019 Apr 30. PMID 31035288
- [Background] Van Regemorter V, Hummel T, Rosenzweig F, Mouraux A, Rombaux P, Huart C. Mechanisms Linking Olfactory Impairment and Risk of Mortality. Front Neurosci. 2020 Feb 21;14:140. doi: 10.3389/fnins.2020.00140. eCollection 2020. PMID 32153360
- [Background] Schambeck SE, Crowell CS, Wagner KI, D'Ippolito E, Burrell T, Mijocevic H, Protzer U, Busch DH, Gerhard M, Poppert H, Beyer H. Phantosmia, Parosmia, and Dysgeusia Are Prolonged and Late-Onset Symptoms of COVID-19. J Clin Med. 2021 Nov 12;10(22):5266. doi: 10.3390/jcm10225266. PMID 34830550
- [Background] Baig AM, Khaleeq A, Ali U, Syeda H. Evidence of the COVID-19 Virus Targeting the CNS: Tissue Distribution, Host-Virus Interaction, and Proposed Neurotropic Mechanisms. ACS Chem Neurosci. 2020 Apr 1;11(7):995-998. doi: 10.1021/acschemneuro.0c00122. Epub 2020 Mar 13. PMID 32167747
- [Background] Meng X, Deng Y, Dai Z, Meng Z. COVID-19 and anosmia: A review based on up-to-date knowledge. Am J Otolaryngol. 2020 Sep-Oct;41(5):102581. doi: 10.1016/j.amjoto.2020.102581. Epub 2020 Jun 2. PMID 32563019
- [Background] Politi LS, Salsano E, Grimaldi M. Magnetic Resonance Imaging Alteration of the Brain in a Patient With Coronavirus Disease 2019 (COVID-19) and Anosmia. JAMA Neurol. 2020 Aug 1;77(8):1028-1029. doi: 10.1001/jamaneurol.2020.2125. No abstract available. PMID 32469400
- [Background] Morbini P, Benazzo M, Verga L, Pagella FG, Mojoli F, Bruno R, Marena C. Ultrastructural Evidence of Direct Viral Damage to the Olfactory Complex in Patients Testing Positive for SARS-CoV-2. JAMA Otolaryngol Head Neck Surg. 2020 Oct 1;146(10):972-973. doi: 10.1001/jamaoto.2020.2366. No abstract available. PMID 32790835
- [Background] Hawkes C. Parosmia: treatment, mechanism, and types. BMJ. 2020 Dec 8;371:m4739. doi: 10.1136/bmj.m4739. No abstract available. PMID 33293264
- [Background] Brann DH, Tsukahara T, Weinreb C, Lipovsek M, Van den Berge K, Gong B, Chance R, Macaulay IC, Chou HJ, Fletcher RB, Das D, Street K, de Bezieux HR, Choi YG, Risso D, Dudoit S, Purdom E, Mill J, Hachem RA, Matsunami H, Logan DW, Goldstein BJ, Grubb MS, Ngai J, Datta SR. Non-neuronal expression of SARS-CoV-2 entry genes in the olfactory system suggests mechanisms underlying COVID-19-associated anosmia. Sci Adv. 2020 Jul 31;6(31):eabc5801. doi: 10.1126/sciadv.abc5801. Epub 2020 Jul 24. PMID 32937591
- [Background] Pace U, Hanski E, Salomon Y, Lancet D. Odorant-sensitive adenylate cyclase may mediate olfactory reception. Nature. 1985 Jul 18-24;316(6025):255-8. doi: 10.1038/316255a0. PMID 3927168
- [Background] Anholt RR. Molecular neurobiology of olfaction. Crit Rev Neurobiol. 1993;7(1):1-22. PMID 8467526
- [Background] Levy LM, Henkin RI, Lin CS, Hutter A, Schellinger D. Increased brain activation in response to odors in patients with hyposmia after theophylline treatment demonstrated by fMRI. J Comput Assist Tomogr. 1998 Sep-Oct;22(5):760-70. doi: 10.1097/00004728-199809000-00019. PMID 9754114
- [Background] Neumann S, Bradke F, Tessier-Lavigne M, Basbaum AI. Regeneration of sensory axons within the injured spinal cord induced by intraganglionic cAMP elevation. Neuron. 2002 Jun 13;34(6):885-93. doi: 10.1016/s0896-6273(02)00702-x. PMID 12086637
- [Background] Moon C, Simpson PJ, Tu Y, Cho H, Ronnett GV. Regulation of intracellular cyclic GMP levels in olfactory sensory neurons. J Neurochem. 2005 Oct;95(1):200-9. doi: 10.1111/j.1471-4159.2005.03356.x. PMID 16181424
- [Background] Henkin RI, Velicu I. cAMP and cGMP in nasal mucus: relationships to taste and smell dysfunction, gender and age. Clin Invest Med. 2008;31(2):E71-7. doi: 10.25011/cim.v31i2.3366. PMID 18377763
- [Background] Henkin RI, Velicu I. cAMP and cGMP in nasal mucus related to severity of smell loss in patients with smell dysfunction. Clin Invest Med. 2008;31(2):E78-84. doi: 10.25011/cim.v31i2.3367. PMID 18377764
- [Background] Henkin RI, Velicu I, Schmidt L. An open-label controlled trial of theophylline for treatment of patients with hyposmia. Am J Med Sci. 2009 Jun;337(6):396-406. doi: 10.1097/MAJ.0b013e3181914a97. PMID 19359985
- [Background] Barnes PJ. Theophylline. Pharmaceuticals (Basel). 2010 Mar 18;3(3):725-747. doi: 10.3390/ph3030725. PMID 27713276
- [Background] Henkin RI, Schultz M, Minnick-Poppe L. Intranasal theophylline treatment of hyposmia and hypogeusia: a pilot study. Arch Otolaryngol Head Neck Surg. 2012 Nov;138(11):1064-70. doi: 10.1001/2013.jamaoto.342. PMID 23165381
- [Background] Goldstein, M.F.; Hilditch, G.J.; Frankel, I.; Chambers, L.; Dvorin, D.J.; Belecanech, G. Intra-nasal theophylline for the treatment of chronic anosmia and hyposmia. Journal of Allergy & Clinical Immunology. 2017;139(2):AB252.
- [Background] Nigwekar SU, Weiser JM, Kalim S, Xu D, Wibecan JL, Dougherty SM, Mercier-Lafond L, Corapi KM, Eneanya ND, Holbrook EH, Brown D, Thadhani RI, Paunescu TG. Characterization and Correction of Olfactory Deficits in Kidney Disease. J Am Soc Nephrol. 2017 Nov;28(11):3395-3403. doi: 10.1681/ASN.2016121308. Epub 2017 Aug 3. PMID 28775001
- [Background] Lee JJ, Peterson AM, Kallogjeri D, Jiramongkolchai P, Kukuljan S, Schneider JS, Klatt-Cromwell CN, Drescher AJ, Brunworth JD, Piccirillo JF. Smell Changes and Efficacy of Nasal Theophylline (SCENT) irrigation: A randomized controlled trial for treatment of post-viral olfactory dysfunction. Am J Otolaryngol. 2022 Mar-Apr;43(2):103299. doi: 10.1016/j.amjoto.2021.103299. Epub 2021 Dec 3. PMID 34894449
- [Background] Lee JJ, Gupta S, Kallogjeri D, Piccirillo JF. Safety of High-Dose Nasal Theophylline Irrigation in the Treatment of Postviral Olfactory Dysfunction: A Dose-Escalation Study. JAMA Otolaryngol Head Neck Surg. 2022 Sep 1;148(9):885-886. doi: 10.1001/jamaoto.2022.1574. PMID 35797023
- [Background] Doty RL, Shaman P, Dann M. Development of the University of Pennsylvania Smell Identification Test: a standardized microencapsulated test of olfactory function. Physiol Behav. 1984 Mar;32(3):489-502. doi: 10.1016/0031-9384(84)90269-5. PMID 6463130
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Busner J, Targum SD. The clinical global impressions scale: applying a research tool in clinical practice. Psychiatry (Edgmont). 2007 Jul;4(7):28-37. PMID 20526405
- [Background] Dunlop BW, Gray J, Rapaport MH. Transdiagnostic Clinical Global Impression Scoring for Routine Clinical Settings. Behav Sci (Basel). 2017 Jun 27;7(3):40. doi: 10.3390/bs7030040. PMID 28653978
- [Background] Mattos JL, Schlosser RJ, Mace JC, Smith TL, Soler ZM. Establishing the minimal clinically important difference for the Questionnaire of Olfactory Disorders. Int Forum Allergy Rhinol. 2018 Sep;8(9):1041-1046. doi: 10.1002/alr.22135. Epub 2018 May 2. PMID 29719139
- [Background] Moscucci M, Byrne L, Weintraub M, Cox C. Blinding, unblinding, and the placebo effect: an analysis of patients' guesses of treatment assignment in a double-blind clinical trial. Clin Pharmacol Ther. 1987 Mar;41(3):259-65. doi: 10.1038/clpt.1987.26. PMID 3816016
- [Background] O'Byrne L, Webster KE, MacKeith S, Philpott C, Hopkins C, Burton MJ. Interventions for the treatment of persistent post-COVID-19 olfactory dysfunction. Cochrane Database Syst Rev. 2021 Jul 22;7(7):CD013876. doi: 10.1002/14651858.CD013876.pub2. PMID 34291813
- [Background] Sorokowska A, Drechsler E, Karwowski M, Hummel T. Effects of olfactory training: a meta-analysis. Rhinology. 2017 Mar 1;55(1):17-26. doi: 10.4193/Rhino16.195. PMID 28040824
- [Background] Whitcroft KL, Hummel T. Clinical Diagnosis and Current Management Strategies for Olfactory Dysfunction: A Review. JAMA Otolaryngol Head Neck Surg. 2019 Sep 1;145(9):846-853. doi: 10.1001/jamaoto.2019.1728. PMID 31318413
- [Background] Nguyen TP, Patel ZM. Budesonide irrigation with olfactory training improves outcomes compared with olfactory training alone in patients with olfactory loss. Int Forum Allergy Rhinol. 2018 Sep;8(9):977-981. doi: 10.1002/alr.22140. Epub 2018 Jun 14. PMID 29901865
- [Background] Tait S, Kallogjeri D, Suko J, Kukuljan S, Schneider J, Piccirillo JF. Effect of Budesonide Added to Large-Volume, Low-pressure Saline Sinus Irrigation for Chronic Rhinosinusitis: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2018 Jul 1;144(7):605-612. doi: 10.1001/jamaoto.2018.0667. PMID 29879268
- [Background] Menorca RM, Fussell TS, Elfar JC. Nerve physiology: mechanisms of injury and recovery. Hand Clin. 2013 Aug;29(3):317-30. doi: 10.1016/j.hcl.2013.04.002. PMID 23895713
- [Background] Wei G, Gu J, Gu Z, Du C, Huang X, Xing H, Li L, Zhang A, Hu X, Huo J. Olfactory Dysfunction in Patients With Coronavirus Disease 2019: A Review. Front Neurol. 2022 Jan 18;12:783249. doi: 10.3389/fneur.2021.783249. eCollection 2021. PMID 35115994
- [Background] Jafar A, Lasso A, Shorr R, Hutton B, Kilty S. Olfactory recovery following infection with COVID-19: A systematic review. PLoS One. 2021 Nov 9;16(11):e0259321. doi: 10.1371/journal.pone.0259321. eCollection 2021. PMID 34752471
- [Derived] Gupta S, Lee JJ, Perrin A, Khan A, Smith HJ, Farrell N, Kallogjeri D, Piccirillo JF. Efficacy and Safety of Saline Nasal Irrigation Plus Theophylline for Treatment of COVID-19-Related Olfactory Dysfunction: The SCENT2 Phase 2 Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2022 Sep 1;148(9):830-837. doi: 10.1001/jamaoto.2022.1573. PMID 35797024

RESULTS

PARTICIPANT FLOW:
Groups:
- Theophylline: 400mg theophylline capsule diluted in 240 mL isotonic nasal saline lavage twice daily.
  Theophylline Powder: Theophylline is a known phosphodiesterase inhibitor in the treatment of asthma. Evidence for post-viral olfactory dysfunction suggests sensory axonal regeneration and olfactory signaling may rely on elevated levels of secondary messengers cAMP and cGMP, a known effect of theophylline. Therefore it is hypothesized to help treat COVID-related smell dysfunction, especially if delivered intranasally.
  Twice daily nasal irrigation with 400 mg theophylline capsules and USP Grade Sodium Chloride & Sodium Bicarbonate Mixture (pH balanced, Isotonic & Preservative & Iodine Free) commercially prepared packets dissolved in 240 ml of distilled water.
- Placebo: 500mg lactose capsule diluted in 240 mL isotonic nasal saline lavage twice daily.
  Theophylline Powder: Theophylline is a known phosphodiesterase inhibitor in the treatment of asthma. Evidence for post-viral olfactory dysfunction suggests sensory axonal regeneration and olfactory signaling may rely on elevated levels of secondary messengers cAMP and cGMP, a known effect of theophylline. Therefore it is hypothesized to help treat COVID-related smell dysfunction, especially if delivered intranasally.
  Twice daily nasal irrigation with 400 mg theophylline capsules and USP Grade Sodium Chloride & Sodium Bicarbonate Mixture (pH balanced, Isotonic & Preservative & Iodine Free) commercially prepared packets dissolved in 240 ml of distilled water.
Period: Overall Study
Arm/Group | Theophylline | Placebo
Started | 26 | 25
Completed | 22 | 23
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Theophylline | Placebo | Total
Number analyzed (Participants) | 26 | 25 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 22 | 47
  >=65 years | 1 | 3 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.43 (11.63) | 47.08 (13.89) | 45.96 (13.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 17 | 36
  Male | 7 | 8 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 26 | 25 | 51

OUTCOME MEASURES:

1. Primary Outcome: UPSIT
Description: UPSIT 0-40 with higher scores indicating better results.
  The response rate defined as the number of participants in each group self-reporting of at least slightly better improvement in the Clinical Global Improvement Scale at 6 weeks post intervention as compared to baseline, devided by the total number of participants in that specific group. The CGI-Improvement Scale has seven response options (from 1 as Very Much Improved to 7 as Very Much Worsened) for answers to the question "Compared to your sense of smell before you started the nasal irrigations, how would you rate your sense of smell now" . Participants reporting 3 as "Minimally Improved", 2 as "Much Improved", or 1 as "Very Much Improved" in the CGI-I will be deemed responders to treatment, and the rate of responders will be compared between the two arms.
Time Frame: Comparison of response rate at 6 weeks post-intervention from baseline between the 2 study groups
Population: This outcome measure could be assessed only from the participants that completed CGI-I at 6 weeks post intervention.
Measure: Number; unit: percentage of participants
Arm/Group | Theophylline | Placebo
Number analyzed (Participants) | 22 | 23
percentage of participants | 59 | 43

2. Secondary Outcome: University of Pennsylvania Smell Identification Test (UPSIT)
Description: UPSIT 0-40 with higher scores indicating better smell.
  This test is an objective, clinically validated 40-question forced-choice odor identification test where microencapsulated odorants on a strip are released by scratching. Out of a total of 40 points, normosmia is defined as ≥34 for males and ≥35 for females, and an increase in ≥4 points will be deemed a clinically significant improvement in symptoms.
Time Frame: Comparison at 6 weeks post-intervention from baseline
Population: The outcome measure could be assessed only on subjects that completed UPSIT test at 6 weeks post-intervention
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Theophylline | Placebo
Number analyzed (Participants) | 22 | 23
score on a scale | 3 [-1 to 7] | 0 [-2 to 6]

3. Secondary Outcome: Change in Questionnaire for Olfactory Dysfunction (QOD) From Baseline to 6 Weeks Post Intervention
Description: Questionnaire for Olfactory Dysfunction (QOD) assesses health-related quality of life of participants based on four factors such as eating, mental health, social interactions, or fear of dysfunction.. The survey also includes questions on parosmia, a phenomena of COVID-related OD. The QOD consists of 17 statements that participants score from 0-3, resulting in a total score from 0 to 51. Higher scores reflect better olfactory-specific QOL.
Time Frame: Comparison at 6 weeks post-intervention from baseline
Population: Since the outcome is measuring the change in QOD, only the data from participant completing QOD at baseline and 6 weeks were included
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Theophylline | Placebo
Number analyzed (Participants) | 22 | 23
score on a scale | 0.86 [-0.57 to 2.85] | 1.43 [-0.29 to 3.14]

4. Secondary Outcome: 36-Item Short Form Health Survey (SF-36)
Description: The SF-36 is a well-established 36-item questionnaire evaluating physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. This test allows us to study the overall quality of life for those suffering from COVID-19 related OD. There is no single overall score for SF-36. The SF 36 generates 8 subscales with scores ranging from 0 (worst) to 100 (best). General health domain scores are reported here.
Time Frame: Baseline assessment
Population: This was a baseline assessment only, so all randomized participants are analyzed.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Theophylline | Placebo
Number analyzed (Participants) | 26 | 25
score on a scale | 75 [40 to 100] | 80 [50 to 100]

5. Secondary Outcome: Olfactory Dysfunction Outcomes Rating (ODOR)
Description: The ODOR is a 28-item QOL instrument with a total score ranging from 0 to 112 points. Higher scores indicate worse QOL with higher degree of dysfunction and limitation. A decrease of 15 or more points is deemed to be a clinically significant improvement in QOL.
Time Frame: Comparison of response rate at 6 weeks post-intervention from baseline between the 2 study groups
Population: This outcome is assessed only for participants that have ODOR assessed at baseline and at 6 months.
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Theophylline | Placebo
Number analyzed (Participants) | 22 | 23
score on a scale | -6.5 [-11.5 to -1.5] | -4.5 [-10.5 to 2]

ADVERSE EVENTS:
Time Frame: All participants were monitored for adverse events throughout participation in the study intervention (week 1 through week 6).
Description: The definition of adverse events/serious adverse events do not differ from the Clinical Trials definition.
Arm/Group | Theophylline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/25
Other Adverse Events (participants affected / at risk) | 7/26 | 11/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Theophylline (N=26) | Placebo (N=25)
fluid retension/extremity swelling (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Event was treated and was defined as mild and not related to study drug
Parosmia and Headache (General disorders) | 1 (1) | 0 (0) — Event was deemed mild and probably related to study drug
Lightheadedness (General disorders) | 2 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (General disorders) | 1 (1) | 2 (2)
Insomnia (General disorders) | 3 (3) | 4 (4)
Tremors (Nervous system disorders) | 2 (2) | 1 (2)
Tachycardia (Cardiac disorders) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-20): https://cdn.clinicaltrials.gov/large-docs/99/NCT04789499/Prot_SAP_000.pdf